CLINICAL TRIAL: NCT06633679
Title: Se Cuida - Internet-delivered Cognitive Behavioral Therapy for Anxiety and Depressive Symptoms in Brazilian Emerging Adults
Brief Title: ICBT for Anxiety and Depressive Symptoms in Brazilian Young Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Gerhard Andersson, PhD, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Se Cuida Brazil
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Anxiety Symptoms; Depressive Symptoms
Keywords: internet-delivered interventions; anxiety; depression; young adults; cognitive-behavioral therapy
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to either intervention or control group. Participants in the control group will receive the same treatment once the intervention group has finished the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Se Cuida Intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Se Cuida Intervention — The intervention consist in an internet based cognitive behavioural therapy program delivered through a online platform. Intervention consist of 8 weeks with 8 weekly modules assigned to the participants. The program has been translated and adapted to the Brazilian and is based on CBT techniques focused on managing psychological symptoms of anxiety and depression in young people. Out of a total 14 modules adaptaded, 8 will be delivered in the treatment: 5 will be available to all participants and 3 will be tailored according to the initial assessment and interviews. The intervention is self-guided with support on demand, meaning that when participants need support, they could chat directly through the platform text message channel with a psychoteraphist responsible for them. Also, once a week each participants receive feedbacks regarding their work on the program's exercises.
  Arms: Intervention group

SUMMARY:
This study aims to investigate the effects of a selfguided internet-based cognitive behavioral therapy (ICBT) program on depressive and anxiety symptoms in young Brazilian adults. Treatment group will be compared to a waiting list control group. Participants will be recruited in Brazil with a nationwide recruitment.

DETAILED DESCRIPTION:
This is a randomized controlled trial carried out to evaluate the effects of an internet-based cognitive behavioral program for depressive and anxiety symptoms in young Brazilians adults. The program consists of 8 weeks of treatment and is carried out through an online platform. During treatment, participants have the support of a therapist who can be reached on demand via the platform's text messaging channel. The program was adapted to Brazilian culture from previous work.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 18 and 24 years old; (2) have a device with Internet access that allows access to the platform; (3) speak and read Brazilian Portuguese.

Exclusion Criteria:

* (1) having a severe psychiatric diagnosis such as bipolar disorder and schizophrenia; (2) having severe suicidal ideation or reported suicidal intent; (3) reporting substance abuse; (4) being in an ongoing psychological and/or psychiatric treatment; (5) changing psychiatric medication less than 3 months before the treatment starts; (6) scoring extremely severe on all three subscales of DASS-21 (28+ for depression, 20+ for anxiety and 34+ for stress.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale - DASS-21 | In recruitment; in every two weeks during treatment; and at the end of treatment after 8 weeks
  Measures depression, anxiety, and stress symptoms in the last week. Primary outcomes will be depressive and anxiety subscales. The instrument consists of 21 questions evaluated with a Likert Scale ranging from 0 (does not apply to me at all) to 3 (applied to me very much or most of the time). The scores for each subscale were proposed by the original authors and range from normal, mild, moderate, severe, and extremely severe symptomatology. The severity rating can be easily accessed in the Brazilian version.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | In recruitment and at the end of treatment after 8 weeks
  Measure sleep problems with 7 questions ranging from 0 to 4 points answers. Symptomatology can vary between non-significant insomnia (0-7), lower limit (8-14), moderate clinical insomnia (15- 21) and severe clinical insomnia (22-28).
Almost Perfect Scale - Revised (APS-R) | In recruitment and at the end of treatment after 8 weeks
  Measures perfectionism symptoms in 23 itens. It has three subscales (Discrepancy, Standards, and Order), with a Likert Scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher values indicate greater perfectionism, with a cut-off score of 42 for the Standards subscale for rating perfectionism. Maladaptive perfectionism is considered if also Discrepancy subscale is 42 or higher.
Brunnsviken Brief Quality of Life Scale (BBQ) | In recruitment and at the end of treatment after 8 weeks
  Measures quality of life with 12 items referring to satisfaction and importance of six areas of life, with responses ranging from 0 (completely disagree) to 5 (completely agree). The scores can range from 0 to 96 points, with a higher score indicating higher quality of life. Clinical populations demonstrated lower scores compared to non-clinical populations, with a mean of 38.7 and 60.1, respectively.
Brazilian adapted version of the Smartphone Addiction Scale-Short Version (SAS-SV) | In recruitment and at the end of treatment after 8 weeks
  Measures problematic Internet use. The scale assesses problematic smartphone use and consists of 33 questions assessed by a Likert Scale ranging from 1 (strongly disagree) to 6 (strongly agree). Problematic use is considered with a cut-off of 31 points for men and 33 for women.
Social Media Disorder Scale-Short Form (SMDS-SF) | In recruitment and at the end of treatment after 8 weeks
  This instrument was translated and adapted for this work. The original scale was developed for adolescents based on the DSM-5 Internet Dependence Disorder criteria and has 9 items assessed by dichotomous yes (1) and no (0) responses. Problematic social media use is considered with a cut-off of 5 points. Additionally, four questions will be included for understanding social medias used, daily usage time, activities performed with social media and primary use.
Depression, Anxiety and Stress Scale - DASS-21 | In recruitment and at the end of treatment after 8 weeks
  Measures depression, anxiety, and stress symptoms in the last week. Stress wil be evaluated as a second outcome. The instrument consists of 21 questions evaluated with a Likert Scale ranging from 0 (does not apply to me at all) to 3 (applied to me very much or most of the time). The scores for each subscale were proposed by the original authors and range from normal, mild, moderate, severe, and extremely severe symptomatology. The severity rating can be easily accessed in the Brazilian version.

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo - Department of Psychology, Faculty of Philosophy, Sciences and Languages of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No